CLINICAL TRIAL: NCT04845685
Title: Hospital Use of CGM (Continuous Glucose Monitor) in Post-operative Patients With Diabetes Mellitus at High Risk for Hypo and Hyperglycemia
Brief Title: A Study to Evaluate Continuous Glucose Monitor in Hospitalized, Post-operative Patients With Diabetes Mellitus
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian G. Dumitrascu, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-010924
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CGM Patients (Experimental): Subjects with diabetes mellitus or medication induced diabetes that have been admitted to the hospital after a surgery for organ transplantation or scheduled for organ transplant surgery will be fitted with a CGM monitor to monitor glucose levels during hospitalization
  Interventions: Device: Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — A device that measures blood sugar levels every 1-5 minutes
  Other Names: Dexcom G6 PRO

SUMMARY:
The purposes of this study is to study if CGMs worn in the postoperative ICU or non-ICU hospital setting have adequate accuracy for blood glucose monitoring when compared to point-of-care (POC) capillary glucometers.

DETAILED DESCRIPTION:
Eligible patients will be approached by research staff either preoperatively or on the first 5 days post-surgery and offered to be enrolled. If agreed to participate, they will be fitted with a blinded CGM monitor (Dexcom G6 PRO) as soon as they are awake and alert after the surgery. They will continue to have their blood glucose check as usual in the ICU and on surgical floors with POC glucometers. On discharge, or at the end of the first CGM sensor life, the sensor will be removed and sensor data will be analyzed. CGM data will be compared with Point-of-Care blood glucose monitoring obtained in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or 2 Diabetes Mellitus.
* Patients 18 years of age or older.
* Admitted for deceased donor renal transplant surgery, pancreas transplant surgery, heart transplant surgery, liver transplant surgery and lung transplant surgery.
* Anticipated minimum of 72h hospital stay.
* Patients on insulin therapy (IV, SQ) post-surgery.

Exclusion Criteria:

* Active COVID-19 infection.
* Pregnant or lactating female.
* Altered Mental Status at the time of sensor placement (sensor will be placed once mental status will improve).
* Inability to provide informed consent.
* Patients taking more than 4 g of acetaminophen in 24 hours or more than 1 gm every 6 hours.

Patients with skin lesions at the application site that may interfere with placement of the sensor.

Patients with known allergy to medical grade adhesive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-12-08 (Estimated); Study Completion 2026-12-08 (Estimated)

PRIMARY OUTCOMES:
CGM accuracy | From date of enrollment and until discharge from the hospital up to 30 days.
  Measured by the mean absolute relative difference (MARD), calculated between matched pairs of POC (point of care) glucose monitors and the closest CGM reading. MARD will be summarized as mean (standard deviation) or median (range) for glucose readings <70g/dl, >180g/dl, >250g/dl respectively.

SECONDARY OUTCOMES:
CGM recorded hypoglycemia episodes | From date of enrollment and until discharge from the hospital up to 30 days.
  The incidence and duration of hypoglycemic episodes
CGM recorded hyperglycemia episodes | From date of enrollment and until discharge from the hospital up to 30 days.
  The incidence of hyperglycemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Dumitrascu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials